CLINICAL TRIAL: NCT01196442
Title: An Expanded Trial of MC5-A Calmare Therapy in the Treatment of Cancer Pain Syndromes and Chronic Chemotherapy-Induced Peripheral Neuropathy Including Pain and Numbness
Brief Title: Electrical Stimulation Pain Therapy in Treating Chronic Pain and Numbness Caused By Chemotherapy in Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-13098; NCI-2010-01945 (Registry Identifier: CTRP)
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Cancer-related Problem/Condition; Neurotoxicity; Pain; Peripheral Neuropathy
MeSH Terms: conditions — Neurotoxicity Syndromes; Pain; Peripheral Nervous System Diseases | interventions — Analgesia; Pain Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I electric stimulation pain therapy (Experimental): Patients undergo electric stimulation pain therapy comprising MC5-A Calmare therapy over 30 minutes once daily for 10 days.
  Interventions: Other: electrical stimulation pain therapy; Other: questionnaire administration

INTERVENTIONS:
Other: electrical stimulation pain therapy — Electrical stimulation pain therapy for 45 minutes on Day 1, then 30 minutes Days 2-10
  Other Names: Calmare; analgesia; cancer pain management; management of cancer pain; pain management; therapy, pain
Other: questionnaire administration — Brief Pain Inventory questionnaire administration at baseline, weekly, then monthly for 3 months

SUMMARY:
RATIONALE: Electrical stimulation pain therapy may help relieve chronic pain and numbness caused by chemotherapy. PURPOSE: This pilot trial studies electrical stimulation pain therapy in treating chronic pain and numbness caused by chemotherapy in patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To evaluate the effect of MC5-A on pain symptoms both immediately and over time.

II. To evaluate the effect of Calmare therapy on other non-pain symptoms. III. To evaluate the effect of MC5-A on daily opioid and other pain medication use.

OUTLINE: Patients undergo electric stimulation pain therapy comprising MC5-A Calmare therapy over 30 minutes once daily for 10 days. After completion of study treatment, patients are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* CIPN neuropathy: received, or currently receiving, neurotoxic chemotherapy (including taxanes-such as paclitaxel or docetaxel, or platinum-based compounds such as carboplatin or cis-platinum or oxaliplatin, or vinca alkaloids such as vincristine, vinblastine, or vinorelbine, or proteosome inhibitors such as bortezomib)
* Pain or symptoms of peripheral neuropathy of >= 1 months duration attributed to chemotherapy-induced peripheral neuropathy
* OR pain of the other types including chemotherapy-induced peripheral neuropathy, numbness predominant; post mastectomy pain; post surgical pain; post herpetic neuropathy; post radiation pain; other (vertebral compression, fracture, miscellaneous)
* The pain must have been stable for at least 2 weeks
* An average daily pain rating of >= 5 out of 10, using the pain numerical rating scale (NRS: 0 is no pain and 10 is worst pain possible); or numbness that bothers the patient at least "a little bit" on the CIPN-20
* Life expectancy >= 3 months
* ECOG performance status 0, 1, or 2

Exclusion Criteria:

* Pregnant women, nursing women, women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, abstinence, etc.)
* Use of an investigational agent for pain control concurrently or =< 30 days
* History of an allergic reaction or previous intolerance to transcutaneous electronic nerve stimulation
* Patients with implantable drug delivery systems, e.g., Medtronic Synchromed
* Patients with heart stents or metal implants such as pacemakers, automatic defibrillators, aneurysm clips, vena cava clips and skull plates (metal implants for orthopedic repair, e.g., pins, clips, plates, cages, joint replacements are allowed)
* Patients with a history of myocardial infarction or ischemic heart disease within the past six months
* Patients with history of epilepsy, brain damage, use of anti-convulsants, symptomatic brain metastases
* Prior celiac plexus block, or other neurolytic pain control treatment within 4 weeks
* Other identified causes of painful paresthesias existing prior to chemotherapy (e.g., radiation or malignant plexopathy, lumbar or cervical radiculopathy, pre-existing peripheral neuropathy of another etiology: B12 deficiency, AIDS, monoclonal gammopathy, diabetes, heavy metal poisoning amyloidosis, syphilis, hyperthyroidism or hypothyroidism, inherited neuropathy)
* Skin conditions such as open sores that would prevent proper application of the electrodes
* Other medical or other condition(s) that in the opinion of the investigators might compromise the objectives of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Swainey, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- See also: VCU Massey Cancer Center — http://www.massey.vcu.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 08/30/2010 through 06/11/2012 at a medical clinical
Pre-assignment Details: No pre-assignment criteria
Groups:
- MC5A Calmare Therapy: Patients undergo electric stimulation pain therapy comprising MC5-A Calmare therapy over 30 minutes once daily for 10 days.
  electrical stimulation pain therapy : Electrical stimulation for 45 minutes on Day 1, then 30 minutes Days 2-10
  questionnaire administration : Brief Pain Inventory at baseline, weekly, then monthly for 3 months
Period: Overall Study
Arm/Group | MC5A Calmare Therapy
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MC5A Calmare Therapy
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 59 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Score From Day 1 to Day 10
Description: Change in Brief Pain Inventory (Now)Scale
  1 (none) to 5 (complete interference)
Time Frame: From day 1 to day 10
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm I: Patients undergo electric stimulation pain therapy comprising MC5-A Calmare therapy over 30 minutes once daily for 10 days.
  Electrical stimulation pain therapy: Electrical stimulation for 45 minutes on Day 1, then 30 minutes Days 2-10
  Questionnaire administration: Brief Pain Inventory at baseline, weekly, then monthly for 3 months
Arm/Group | Arm I
Number analyzed (Participants) | 39
units on a scale | -3.3 (0.7)

2. Secondary Outcome: Effect of Electrical Stimulation Pain Therapy on Other Non-pain Symptoms at Day 1
Description: Chemotherapy-induced peripheral neuropathy (CIPN)-20. The CIPN-20 has 3 subscales: a sensory, motor, and autonomic subscale. There are 17 questions that are rated 0-not at all to 3-very much. Scales are summed. Final score ranges from 0-51, 0 as the best possible outcome and 51 as the worst.
Time Frame: Day 1
Population: Participants at Day 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | MC5A Calmare Therapy
Number analyzed (Participants) | 39
units on a scale
  sensory symptoms | 20.4129 (0.9114)
  motor symptoms | 15.6268 (0.7598)

3. Secondary Outcome: Use of Medications Including Morphine Oral Dose Equivalents, Anti-depressants, and Neuroleptics
Description: Record daily pain medication usage and convert all opioids to MOEDs (American Pain Society 2003). Compare the average daily use prior to day 1 to the average daily use day 30. Range is 0-none to 240-most
Time Frame: From day 1 to day 30
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | MC5A Calmare Therapy
Number analyzed (Participants) | 39
doses | 28.9 (47.3)

4. Secondary Outcome: Effect of Electric Stimulation Pain Therapy on Other Non-pain Symptoms at Day 10
Description: as for outcome 2
Time Frame: Day 10
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | MC5A Calmare Therapy
Number analyzed (Participants) | 33
units on a scale
  sensory symptoms | 17.8305 (0.9437)
  motor symptoms | 14.1815 (0.7878)

5. Secondary Outcome: Effect of Electric Stimulation Pain Therapy on Other Non-pain Symptoms at Month 1
Description: as for outcome 2
Time Frame: month 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | MC5A Calmare Therapy
Number analyzed (Participants) | 33
units on a scale
  snesory symptoms | 16.5207 (0.9345)
  motor symptoms | 13.5443 (0.7797)

6. Secondary Outcome: Effect of Electric Stimulation Pain Therapy n Other Non-pain Symptoms at Month 2
Description: as for outcome 2
Time Frame: month 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | MC5A Calmare Therapy
Number analyzed (Participants) | 32
units on a scale
  sensory symptoms | 16.4723 (0.9480)
  motor symptoms | 13.3816 (0.7917)

7. Secondary Outcome: Effect of Electric Stimulation Pain Therapy on Other Non-pain Symptoms at Month 3
Description: as for outcome 2
Time Frame: Month 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | MC5A Calmare Therapy
Number analyzed (Participants) | 32
units on a scale
  sensory symptoms | 17.3325 (0.9388)
  motor symptoms | 12.8499 (0.7835)

ADVERSE EVENTS:
Time Frame: While patients are active in trial: During 10 days of treatment and followed for 3 months after treatment.
Arm/Group | MC5A Calmare Therapy
Serious Adverse Events (participants affected / at risk) | 1/39
Other Adverse Events (participants affected / at risk) | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MC5A Calmare Therapy (N=39)
Thromboembolic event (Vascular disorders) | 1 (1) — Unrelated (Grade 2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No